CLINICAL TRIAL: NCT05967910
Title: The Effect of Chronic Stress on Efficacy of Immune Checkpoint Inhibitors in Patients With Newly Diagnosed Esophageal Cancer
Brief Title: The Effect of Chronic Stress on Efficacy of ICIs in Esophageal Cancer Patients (STRESS-ESCA Study)
Acronym: STRESS-ESCA
Status: Recruiting | Type: Observational
Sponsor: Second Xiangya Hospital of Central South University (Other)
Collaborators: The First Affiliated Hospital of Hunan University of Traditional Chinese Medicine (Other); Changsha Central Hospital (Other)
Responsible Party: Principal Investigator, Fang Wu, chief physician, Second Xiangya Hospital of Central South University
Other Study IDs: XYEYY2023052602
Record Dates: First submitted 2023-05-24; First posted 2023-08-01 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Esophageal Cancer; Immunotherapy
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Early esophageal cancer patients with chronic psychological stress
  Interventions: Other: chronic psychological stress
- Early esophageal cancer patients without chronic psychological stress
- Advanced esophageal cancer patients with chronic psychological stress
  Interventions: Other: chronic psychological stress
- Advanced esophageal cancer patients without chronic psychological stress

INTERVENTIONS:
Other: chronic psychological stress — Chronic psychological stress includes symptoms of anxiety and depression.
  Groups: Advanced esophageal cancer patients with chronic psychological stress; Early esophageal cancer patients with chronic psychological stress

SUMMARY:
Chronic stress refers to a special emotional state caused by unexpected stress for a long time, with an increasing incidence in the population. It can cause the body to release hormones such as cortisol and adrenaline. Tumor patients often experience changes such as psychological and emotional abnormalities, decreased quality of life, and impaired social relationships. Under stimulation, patients often experience negative reactions such as anxiety or depression. Epidemiological studies have shown that stress can affect the prognosis of malignant tumors, but the effect of stress on the efficacy and prognosis of esophageal cancer is still unclear.

In animal models, chronic stress leads to an increase in tissue catecholamine levels, increased tumor burden, and increased invasiveness of ovarian cancer cells in mouse models. At the same time, stress can promote tumor neovascularization in mice. However, the mechanism by which chronic stress affects the occurrence and development of esophageal cancer is currently unclear. In addition to neurohumoral factors, chronic stress can cause changes in the gut microbiota, which in turn affects the body's digestion, metabolism, and immune function. It is a key gatekeeper of the immune response to tumors. Therefore, gut microbiota as an intermediate factor may also affect the occurrence and prognosis of various types of esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤ 75 years old
2. Pathologically diagnosed as esophageal cancer
3. Patient tumor tissue samples can be obtained
4. At least one measurable lesion can be evaluated according to the RECIST 1.1 standard
5. As a newly treated patient, they have not received systematic anti-tumor treatment for locally advanced or metastatic chest tumors
6. There is no obvious abnormality in the electrocardiogram and no obvious cardiac dysfunction
7. Hematology and liver and kidney function indicators meet the requirements

Exclusion Criteria:

1. Merge with other malignant tumors
2. Long term use of hormones or immunosuppressants
3. Concomitant acute or chronic mental illness
4. Patients who have been taking drugs that can alter the activity of the sympathetic nervous system for a long time or are currently taking them
5. Other malignant diseases that require systematic treatment
6. Patients who have undergone other clinical drug experiments before
7. Patients with symptomatic brain metastases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 cases of esophageal cancer patient are required and is divided into two groups: the experimental group (stress group) and the control group (non stress group) within each early and late stage group.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 3 years
  The proportion of patients with a complete response or partial response to treatment according to Response Evaluation Criteria in Solid Tumors (RECIST v1.1)
Progression-free survival (PFS) | 3 years
  Time from the beginning of first-line immunotherapy to the first progression(PD) in patients with advanced esophageal cancer
Effect of Chronic stress on efficacy of immune checkpoint inhibitors | 3 years
  The chronic stress status including depression and anxiety symptoms.We will use two types of questionnaires, Patient Health Questionnaire-9 (PHQ-9) and Generalized Anxiety Disorder-7 (GAD-7), as a whole to conduct a comprehensive psychological assessment of patients. And then evaluate the impact of chronic stress status on the efficacy of immune checkpoint inhibitors, including ORR, PFS, and OS.
  PHQ-9 has 9 items, each on a scale of 0 to 3. The sum score (range 0 to 27) indicates the degree of depression, with scores of 5, 10, 15, and 20 represent mild, moderate, moderate to severe and severe levels of depression.
  GAD-7 has 7 items, each on a scale of 0 to 3. Higher total scores (ranging from 0 to 21) indicate higher anxious symptoms with 5 to 9 classified as mild, 10 to 14 classified as moderate, and 15 to 21 classified as moderate-severe.

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years
  Overall survival (OS) is defined as the duration from the beginning of first-line immunotherapy until death due to any cause. Subjects who are still alive at the end of the study observation period will be censored at the time of last known vital status.
Effect of chronic stress on quality of life | 5 years
  Chronic stress status including depression and anxiety symptoms.We will use Short Form Health Survey 36 (SF-36) and EORTC QLQ-C30 (version. 3) questionnaires as a whole to evaluate the quality of life of patients.
  SF-36 includes 36 items and assesses the functional status and well-being on eight multi-item subscales. The total score on each SF-36 subscale ranges between 0 and 100. A greater score indicates better QoL.
  The EORTC QLQ-C30 is composed of 9 multi-item scales: 5 functioning scales (physical, role, cognitive, emotional, and social), a global QOL scale, and 3 symptom scales (fatigue, pain, and nausea/vomiting). All scales and single items are linearly transformed to an 0-100 scale. A higher score represents a better level of functioning.

OTHER OUTCOMES:
The correlation between gut microbiota and chronic stress and the efficacy of ICIs | 5 years
  The baseline fetal is collected and assessed by 16S rRNA sequencing. We will measure the abundance of gut microbiota such as Bacteroides, Lactobacillus, and Ackermann's bacteria through 16s RNA sequencing. And expose the association between gut microbiota and chronic stress (PHQ-9 and GAD-7) and the efficacy of ICIs (ORR, PFS, and OS) during the enrolled observation process through correlation analysis.
The correlation between tumor microenvironment signature and chronic stress and the efficacy of ICIs | 5 years
  The baseline paraffin-embedded tissue is collected and assessed by multiplex immunohistochemistry, including T lymphocytes, B lymphocytes, NK lymphocytes, macrophagocyte, and DC cells. And explore the association between tumor microenvironment signature and chronic stress (PHQ-9 and GAD-7) and the efficacy of ICIs (ORR, PFS, and OS) during the enrolled observation process through correlation analysis.
The correlation between peripheral immune cells signature and chronic stress and the efficacy of ICIs | 5 years
  The baseline peripheral venous blood is collected and assessed by flow cytometry, including T lymphocytes, B lymphocytes, NK lymphocytes, macrophagocyte, and DC cells. And explore the association between peripheral immune cells signature signature and chronic stress (PHQ-9 and GAD-7) and the efficacy of ICIs (ORR, PFS, and OS) during the enrolled observation process through correlation analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oncology, The Second Xiangya Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No